CLINICAL TRIAL: NCT04039594
Title: Outcomes of Patients With Venoarterial Extracorporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Chief, Center for Cardiac Intensive Care, Beijing Anzhen Hospital
Other Study IDs: 2019027X
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Cardiogenic Shock; Cardiac Arrest
Keywords: extracorporeal life support, extracorporeal membrane oxygenation, cardiogenic shock, cardiac arrest
MeSH Terms: conditions — Shock, Cardiogenic; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO
  Interventions: Device: VA ECMO

INTERVENTIONS:
Device: VA ECMO — VA ECMO for cardiopulmonary support

SUMMARY:
Venoarterial extracorporeal membrane oxygenation (VA ECMO)-also referred to as extracorporeal life support-is a form of temporary mechanical circulatory support and simultaneous extracorporeal gas exchange. The objective of this observational, cohort study is to evaluate the short-term and long-term outcomes of patients with VA ECMO.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving VA ECMO for cardiopulmonary support

Exclusion Criteria:

Refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving VA ECMO for cardiopulmonary support
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 365 days
Rate of successful weaning from ECMO | 30 days
ECMO-related complications | 30 days
  Bleeding requiring transfusion or surgery, stroke, sepsis, limb ischemia requiring intervention, system or cannula change
Other complications | 30 days
  Acute renal failure, ulcer bleeding, pneumonia, sepsis
Duration stay at ICU and hospital | 365 days

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China